CLINICAL TRIAL: NCT03697434
Title: Pilot to Assess the Acceptance of Palliative Care Referral Among Those With Parkinson Disease
Brief Title: Acceptability of Palliative Care in Parkinson Disease Care
Acronym: Palliate-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: American Academy of Neurology (Other)
Responsible Party: Principal Investigator, Christopher Tarolli, Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 72429
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Palliative Care referral (Experimental): Participants with specific uncontrolled symptoms or critical events in course of their Parkinson disease will be referred to a palliative care specialist for supportive care.
  Interventions: Behavioral: Palliative Care referral

INTERVENTIONS:
Behavioral: Palliative Care referral — Individuals with Parkinson disease identified as having specific uncontrolled symptoms or critical events will undergo standardized referral to palliative care, who will provide supportive care. During the palliative care referral, participants and their care partners may discuss symptoms, disease burden (physical, emotion, financial, and psychological), quality of life, goals of care, and advance directive completion. Palliative care specialists may recommend interventions to manage bothersome symptoms or to improve disease burden for both participants and care partners.

SUMMARY:
This study will assess the feasibility of using specific criteria to standardize the referral of individuals with Parkinson disease to a group of medical providers known as palliative care specialists. Palliative care specialists provide supportive care to individuals living with serious illnesses. The specialty focuses on providing relief from the symptoms and stress of serious illness.

ELIGIBILITY:
Subjects with Parkinson disease:

Inclusion Criteria:

* Diagnosis of idiopathic PD confirmed as most likely diagnosis with participant's treating provider
* 18 years of age or older
* Participant or care partner able to provide informed consent
* Presence of one or more of the following:

Uncontrolled symptoms (over prior week):

* Depression
* Pain
* Fatigue

Critical events (over prior 6 months):

* ≥3 falls
* Unintended weight loss
* Wheelchair dependence (>50% of time)

Exclusion Criteria:

* Diagnosis of atypical or secondary parkinsonism
* Outpatient palliative care visit scheduled or within the prior 6 months of the screening visit

Subjects who are care partners:

Inclusion Criteria:

* Care partner of enrolled participant in the study
* 18 years of age or older
* Able to provide informed consent

Exclusion Criteria:

• No care partner specific exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-02 (Actual)

PRIMARY OUTCOMES:
Proportion of enrolled participants who have at least 1 visit with a palliative care provider within 3 months of referral | 3 months
  We will assess the feasibility of standardized referral to palliative care by calculating the proportion of enrolled participants with Parkinson disease who have at least 1 visit with a palliative care provider within 3 months of referral.

SECONDARY OUTCOMES:
Change in mean symptom burden | Baseline to 3 months
  Symptom burden will be measured using the Edmonton Symptom Assessment Scale-Revised for Parkinson Disease (ESAS-R: PD), which measures the severity of 14 symptoms on a 1-10 scale. Scores range from 0-140 with higher scores indicating higher symptom burden.
Change in mean quality of life as assessed by the Quality of Life-Alzheimer Disease questionnaire (QoL-AD) | Baseline to 3 months
  Quality of life will be measured using the Quality of Life-Alzheimer Disease questionnaire, which is a 13-item measure that assesses overall quality of life with a focus on physical, social, psychological, and spiritual well-being. Scores range from 13-52 with higher scores indicating better quality of life.
Change in mean caregiver burden | Baseline to 3 months
  Caregiver burden will be measured using the Zarit Burden interview, which is a 22-item questionnaire that assesses caregiver fear, anger, guilt, perspective, hope, and overall quality of life. Scores range from 0-88 with a score of 0-21 associated with little or no burden, 21-40 mild to moderate burden, 41-60 moderate to severe burden, and 61-88 severe burden.
Change in mean caregiver self-efficacy | Baseline to 3 months
  Caregiver self-efficacy will be measured using the Revised Scale for Caregiver Self-efficacy, which is a 15-item questionnaire with 3 sub-sections (self-efficacy for obtaining respite, self-efficacy for responding to disruptive patient behaviors, and self-efficacy for controlling upsetting thoughts about caregiving). Respondents rate their certainty of being able to complete each task from 0% (cannot perform task at all) to 100% (certain that task can be performed). Scores on each of the sub-sections range from 0-500 with a higher score indicating greater self-efficacy.
Barriers to palliative care referral | Baseline
  Barriers to palliative care referral will be measured using a novel qualitative survey that assesses perceived barriers to referral and drivers of desire for referral to palliative care among those with Parkinson disease. The measure includes a qualitative survey of 9 potential barriers to consultation and 5 potential reasons to undergo consultation. Respondents can select as many barriers or reasons as applicable to their perception of referral and can provide free text responses. Overall frequency of selection of each identified barrier among participants will be assessed both at baseline and at 3 months following palliative care referral. Barriers and reasons for referral with higher frequency will be considered to be more important in hindering or driving desire for referral, respectively.
Barriers to palliative care referral | 3 months
  Barriers to palliative care referral will be measured using a novel qualitative survey that assesses perceived barriers to referral and drivers of desire for referral to palliative care among those with Parkinson disease. The measure includes a qualitative survey of 9 potential barriers to consultation and 5 potential reasons to undergo consultation. Respondents can select as many barriers or reasons as applicable to their perception of referral and can provide free text responses. Overall frequency of selection of each identified barrier among participants will be assessed both at baseline and at 3 months following palliative care referral. Barriers and reasons for referral with higher frequency will be considered to be more important in hindering or driving desire for referral, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- URMC Neurology; 919 Westfall Rd, Building C, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No